CLINICAL TRIAL: NCT01756079
Title: A Multi-centre Single-arm Study to Evaluate the Efficacy and Safety of BOCEPREVIR 44 Weeks in Addition to Standard of Care (SOC) in Previously Treatment Failure (Relapser, Non-responders, Both Partial and Null) Patients With Chronic Hepatitis C Genotype 1 (G1) and Cirrhosis (F4 Metavir). (MK-3034-105)
Brief Title: A Study to Evaluate the Efficacy and Safety of Boceprevir Added to Standard of Care Therapy in Previously Treated Participants With Chronic Hepatitis C Genotype 1 and Cirrhosis (MK-3034-105)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3034-105; 2012-002772-13 (EudraCT Number)
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PegIFN-2b + RBV+ boceprevir (Experimental): Participants will receive PegIFN-2b (once weekly, 1.5 µg/kg subcutaneously) + RBV (capsules, orally, weight-based dose from 800-1400 mg/day divided into two daily doses) for 4 weeks and then will receive 44 additional weeks of treatment with PegIFN-2b (once weekly, 1.5 µg/kg subcutaneously) + RBV (capsules, orally, weight-based dose from 800-1400 mg/day divided into two daily doses) + boceprevir (capsules, orally, 800 mg three times per day).
  Interventions: Drug: boceprevir; Biological: PegIFN-2b; Drug: RBV

INTERVENTIONS:
Drug: boceprevir
  Other Names: SCH 503034
Biological: PegIFN-2b
  Other Names: Peginterferon alfa-2b; PegIntron; SCH 054031
Drug: RBV
  Other Names: Ribavirin; Rebetol

SUMMARY:
This study is being done to find out if the addition of boceprevir to standard of care (SOC) treatment with peginterferon alfa-2b (PegIFN-2b) + ribavirin (RBV) is effective for participants with chronic hepatitis C (CHC) genotype 1 and cirrhosis who were not successfully treated by previous SOC. All participants will receive treatment with SOC alone for 4 weeks and then boceprevir will be added to the treatment regimen for 44 additional weeks of combined treatment.

ELIGIBILITY:
Inclusion criteria:

* Weight between 40 kg and 125 kg
* Documented CHC genotype 1 infection
* Previous course of treatment with SOC (PegIFN-2a or PegIFN-2b + RBV) with a documented non-response
* Documented diagnosis of cirrhosis
* No evidence of hepatocellular carcinoma (HCC) by ultrasound
* Participant and partner of participant must agree to use 2 effective contraceptives as specified for at least 2 weeks prior to Day 1 of treatment and continue until at least 6 months after last dose of study drug (7 months for male participants)

Exclusion criteria:

* Co-infection with human immunodeficiency virus (HIV) or hepatitis B virus
* Use of any investigational drugs within 30 days prior to study enrollment
* Participation in any other clinical trial within 30 days of study enrollment or intention to participate in another clinical trial during this study
* Evidence of present or previous decompensated liver disease including, but not limited to, a history or presence of clinical ascites or hepatic encephalopathy. Only participants with large (F3) esophageal varices, as determined in an esophagogastroduodenoscopy (EGD) performed within the past 12 months according to international guidelines will be excluded.
* Clinically significant ocular examination findings
* Pre-existing significant psychiatric condition(s)
* Clinical diagnosis of active or recent substance abuse
* Evidence of active or suspected malignancy, or a history of malignancy, within the last 3 years (except adequately treated carcinoma in situ and basal cell carcinoma of the skin)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-02-06 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 130 participants were screened. Sixty participants passed screening, but 2 of these participants were excluded before assignment because standard of care treatment was not received during the Lead-in Period.
Groups:
- Overall Participants: Participants received PegIFN-2b (once weekly, 1.5 µg/kg subcutaneously) + RBV (capsules, orally, weight-based dose from 800-1400 mg/day divided into two daily doses) for 4 weeks during the Lead-in Period and then 44 additional weeks of treatment in the Treatment Period receiving PegIFN-2b (once weekly, 1.5 µg/kg subcutaneously) + RBV (capsules, orally, weight-based dose from 800-1400 mg/day divided into two daily doses) + boceprevir (capsules, orally, 800 mg three times per day). After completion of treatment, follow-up continued for an additional 24 weeks.
Period: Lead-in: Day 0 to Week 4
Arm/Group | Overall Participants
Started | 58
Completed | 58
Not Completed | 0
Period: Treatment / Follow-up: Week 4 to Week 72
Arm/Group | Overall Participants
Started | 58
Treated in Treatment Period | 54
Completed | 23
Not Completed | 35
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 5
Not completed — No information available | 2
Not completed — Lack of Efficacy | 20
Not completed — No boceprevir during Treatment Period | 4

BASELINE CHARACTERISTICS:
Population: All participants who received PegIFN-2b + RBV during the Lead-in Period
Arm/Group | Overall Participants
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Sustained Virological Response at Follow-up Week 24 (SVR24)
Description: Hepatitis C Virus (HCV) ribonucleic acid (RNA) was measured using a polymerase chain reaction assay. SVR24 was defined as HCV RNA less than the Limit of Quantification (<25 International Units (IU)/mL) 24 weeks after the end of the Treatment Period.
Time Frame: Week 72 (24 weeks after end of treatment)
Population: The Intent to Treat population included all participants who received at least 1 administration of boceprevir during the Treatment Period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 54
Percentage of participants | 35.2 [22.7 to 49.4]

2. Primary Outcome: Percentage of Participants With One or More Adverse Events
Description: Adverse events were monitored during the Lead-in and Treatment Periods
Time Frame: Up to 48 weeks (Lead-in and Treatment Periods)
Population: Safety Analysis Set 2 included all participants who received boceprevir during the Treatment Period
Measure: Number; unit: Percentage of participants
Groups:
- Overall Participants: Participants received PegIFN-2b (once weekly, 1.5 µg/kg subcutaneously) + RBV (capsules, orally, weight-based dose from 800-1400 mg/day divided into two daily doses) for 4 weeks during the Lead-in Period and then 44 additional weeks of treatment in the Treatment Period receiving PegIFN-2b (once weekly, 1.5 µg/kg subcutaneously) + RBV (capsules, orally, weight-based dose from 800-1400 mg/day divided into two daily doses) + boceprevir (capsules, orally, 800 mg three times per day).
Arm/Group | Overall Participants
Number analyzed (Participants) | 54
Percentage of participants | 98.1

3. Primary Outcome: Percentage of Participants With an Adverse Event Leading to Discontinuation of Study Medication
Description: Adverse events were monitored during the Lead-in and Treatment Periods
Time Frame: Up to 48 weeks (Lead-in and Treatment Periods)
Population: Safety Analysis Set 2 included all participants who received boceprevir during the Treatment Period
Measure: Number; unit: Percentage of participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 54
Percentage of participants | 9.3

ADVERSE EVENTS:
Time Frame: Up to 72 weeks (including Lead-in, Treatment, and Follow-up Periods)
Description: Safety Analysis Set 1 included all participants who received PegIFN-2b + RBV during the Lead-in Period
Groups:
- Overall Participants: Lead-in, Treatment and Follow-up: Participants received PegIFN-2b (once weekly, 1.5 µg/kg subcutaneously) + RBV (capsules, orally, weight-based dose from 800-1400 mg/day divided into two daily doses) for 4 weeks during the Lead-in Period and then 44 additional weeks of treatment in the Treatment Period receiving PegIFN-2b (once weekly, 1.5 µg/kg subcutaneously) + RBV (capsules, orally, weight-based dose from 800-1400 mg/day divided into two daily doses) + boceprevir (capsules, orally, 800 mg three times per day). After completion of treatment, follow-up continued for an additional 24 weeks.
Arm/Group | Overall Participants: Lead-in, Treatment and Follow-up
Serious Adverse Events (participants affected / at risk) | 10/58
Other Adverse Events (participants affected / at risk) | 56/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Participants: Lead-in, Treatment and Follow-up (N=58)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Hyperpyrexia (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Parathyroid fever (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Participants: Lead-in, Treatment and Follow-up (N=58)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 44 (82)
Nausea (Gastrointestinal disorders) | 12 (13)
Adverse drug reaction (General disorders) | 11 (11)
Asthenia (General disorders) | 35 (42)
Influenza like illness (General disorders) | 5 (12)
Pyrexia (General disorders) | 15 (35)
Accidental overdose (Injury, poisoning and procedural complications) | 5 (5)
Headache (Nervous system disorders) | 6 (8)
Leukopenia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 16 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 6 (10)
Decreased appetite (Metabolism and nutrition disorders) | 12 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 14 (15)
Syncope (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 7 (7)
Irritability (Psychiatric disorders) | 3 (3)
Nocturia (Renal and urinary disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 7 (9)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Lacrimation increased (Eye disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.